CLINICAL TRIAL: NCT00009217
Title: Treatment of Behavioral Symptoms in Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #4051R; R01MH055735 (NIH); NCT00000183 (obsolete NCT alias)
Record Dates: First submitted 2001-01-23; First posted 2001-01-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2012-02

CONDITIONS: Alzheimer's Disease; Psychosis; Agitation
Keywords: Alzheimer's disease; psychosis; agitation; haloperidol
MeSH Terms: conditions — Alzheimer Disease; Psychotic Disorders; Psychomotor Agitation | interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haloperidol-Haloperidol (Active Comparator): Haloperidol for 20 weeks followed by haloperidol for 24 weeks
  Interventions: Drug: Haloperidol-Haloperidol
- Haloperidol-Placebo (Placebo Comparator): Haloperidol for 20 weeks followed by placebo for 24 weeks
  Interventions: Drug: Haloperidol-Placebo

INTERVENTIONS:
Drug: Haloperidol-Haloperidol — Haloperidol open label flexible dose 1-5 mg daily for 20 weeks followed by haloperidol double-blind 1-5 mg for 24 weeks
  Other Names: Haldol
  Arms: Haloperidol-Haloperidol
Drug: Haloperidol-Placebo — Haloperidol open-label flexible dose of 1-5 mg for 20 weeks followed by placebo double-blind for 24 weeks
  Other Names: Haldol
  Arms: Haloperidol-Placebo

SUMMARY:
The optimal strategy for the treatment of behavioral complications in patients with probable Alzheimer's disease (AD) remains unclear.

The objective of this study is to evaluate the risk of relapse following discontinuation of haloperidol in patients with Alzheimer's disease (AD) with psychosis or agitation who respond to it.

In Phase A of this study, AD outpatients with behavioral complications receive 20 weeks of open haloperidol treatment with an oral dose of 1-5 mg daily, titrated individually to achieve the optimal trade-off between efficacy and side effects. Responders to Phase A participate in Phase B, a 24-week continuation trial in which patients are randomized to continuation haloperidol or placebo.

The primary outcome is the time to relapse of psychosis or behavioral disturbance.

DETAILED DESCRIPTION:
The study involves two phases. Outpatients with AD who meet inclusion/ exclusion criteria enter Phase A, the 20 week open acute treatment phase that uses a flexible dose regimen of haloperidol 1-5 mg daily. Haloperidol is started at an oral dose of 1 mg daily, with subsequent dose titration in 1 mg increments until the optimal dose is reached, i.e., optimal trade-off between efficacy and side effects. At the end of Phase A, patients who do not meet criteria for clinical response exit the protocol and is treated openly with alternative medications.

Phase A responders enter Phase B, a 24-week random assignment, placebo-controlled, continuation trial. Randomization is stratified by the severity of dementia and by the presence of psychosis. Half the patients are randomized to haloperidol (continuing at the same dose as at the end of Phase A), and the other half are randomized to placebo. Patients who relapse during Phase B exit the protocol and receive open treatment.

In Phase A, patients are followed at 0, 2, 4 weeks and every 4 weeks thereafter until 20 weeks. In the discontinuation trial, Phase B, patients are followed at 0, 1, 2, 4, week time points and every 4 weeks thereafter until 24 weeks. If a patient shows signs of relapse, the patient is brought in for more frequent visits, regardless of the stage of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for dementia either sex, age 50-95 years
* Meets NINCDS-ADRDA criteria for probable Alzheimer's disease
* Meets Folstein Mini-Mental State Exam score of 5-26, inclusive
* Intellectual impairment reported for at least six months
* Availability of family member who has had direct contact with the patient for an average of at least once every week during the three months prior to study entry
* Has current symptoms of psychosis or agitation. Criteria for "psychosis" requires the presence of delusions and/or hallucinations identified by the Columbia University Scale for Psychopathology in Alzheimer's Disease (CUSPAD) and a minimum Brief Psychiatric Rating Scale (BPRS) psychosis factor score of at least 4 (moderate severity) on one of the following two items: These two items comprise the psychosis factor, excluding the item for conceptual disorganization. Agitation is defined as a score of greater than 3 (present at least 10 days per month) on one or more of the CERAD Behavioral Rating Scale for Dementia items for agitation, purposeless wandering, verbal aggression or physical aggression.
* Free of psychotropic medication for at least two weeks prior to study entry, or able to tolerate medication washout for this period.
* Informed consent by patient and family member, as per IRB procedures at New York State Psychiatric Institute.

Exclusion Criteria:

* Acute unstable medical condition, delirium, alcohol or substance abuse or dependence within the past 1 year
* Clinical evidence of stroke, other dementias including vascular or Lewy body or frontotemporal dementia, multiple sclerosis, Parkinson's disease, Huntington's disease, tardive dyskinesia
* Diagnosis of a psychotic disorder antedating the onset of dementia
* Antipsychotic medication usage during 4 weeks prior to study entry
* Contraindication to the use of haloperidol

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 1999-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
For the primary hypothesis, the primary endpoint is time to relapse. | 0-24 weeks in Phase B

SECONDARY OUTCOMES:
Severity of target symptoms at the end of Phase A as a predictor of relapse | 0-24 weeks in Phase B
Severity of Brief Psychiatric Rating Scale psychosis and hostile suspiciousness factor scores | 0-20 weeks in Phase A and 0-24 weeks in Phase B
MMSE and Blessed Functional Activity Scale | 0-20 weeks in Phase A and 0-24 weeks in Phase B

CONTACTS AND LOCATIONS:
Overall Officials: Davangere Devanand, M.D., Principal Investigator — Columbia University College of Physicians and Surgeon
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Result] Devanand DP, Pelton GH, Cunqueiro K, Sackeim HA, Marder K. A 6-month, randomized, double-blind, placebo-controlled pilot discontinuation trial following response to haloperidol treatment of psychosis and agitation in Alzheimer's disease. Int J Geriatr Psychiatry. 2011 Sep;26(9):937-43. doi: 10.1002/gps.2630. Epub 2010 Dec 28. PMID 21845596
- See also: link to Pubmed abstract — http://www.ncbi.nlm.nih.gov/pubmed/21845596